CLINICAL TRIAL: NCT00219349
Title: Cognitive-Behavioral Therapy and Pharmacotherapy Augmentation for Generalized Anxiety Disorder: A Pilot Investigation
Brief Title: Cognitive-Behavioral Therapy and Escitalopram for Generalized Anxiety Disorder(GAD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #4941
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Results first posted 2012-05-09 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: Generalized Anxiety Disorder
Keywords: Anxiety Disorders; Anxiety Neuroses; Behavior Therapy, Cognitive; Escitalopram
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — Cognitive Behavioral Therapy; Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Escitalopram (Experimental): 12 weeks of open label escitalopram, 10-20 mg/day (after 14 weeks of cognitive behavioral therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy; Drug: escitalopram

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — 14 weekly sessions of individualized CBT
Drug: escitalopram — 10-20 mg per day for 12 weeks
  Other Names: lexapro

SUMMARY:
The goals of this pilot study are as follows:

1) To disseminate and examine the effectiveness of a manualized, individual, cognitive-behavioral psychotherapy (CBT) for adults with Generalized Anxiety Disorder(GAD), 2) to test the effectiveness of augmentation (the addition of) antidepressant therapy in participants who do not fully respond to CBT, and 3) to examine individual and clinical predictors of non-response to CBT and predictors of response to augmentation antidepressant therapy. A related goal is to examine the maintenance of treatment gains obtained from CBT alone and CBT with augmentation antidepressant therapy, over a twenty-four month follow-up period. This study will serve as a pilot investigation in preparation for a larger federally funded study using this treatment approach. We hypothesize that CBT will result in remission (no longer having GAD) and/or high endstate functioning (clinically meaningful improvement) in approximately 40-50% of participants. Further, we hypothesize that augmentation antidepressant therapy in participants who do not fully respond to CBT will result in further clinically significant improvement.

DETAILED DESCRIPTION:
This pilot investigation will examine the effectiveness of augmenting cognitive behavioral therapy (CBT) with antidepressant pharmacotherapy (escitalopram[Lexapro]) in adults with generalized anxiety disorder (GAD) who do not fully respond to a temporally primary trial of CBT. A secondary aim of this study is to assess the maintenance of treatment gains made by patients in response to CBT, and to CBT with antidepressant augmentation therapy, over a two-year follow-up period.

CBT is an empirically supported psychotherapy that has been found to be effective in treating GAD in approximately 50 percent of patients enrolled in controlled clinical trials. However, a substantial proportion (nearly half) of individuals with GAD do not achieve full remission or clinically significant improvement at the cessation of CBT. Escitalopram (Lexapro)is a selective serotonin reuptake inhibitor (SSRI) antidepressant, which has been shown to be effective in treating GAD in several large-scale controlled clinical trials. The Food and Drug Administration has approved ecitalopram for the treatment of GAD.

The proposed research plan encompasses the conduct of an open clinical trial (No randomized placebo control) of 14 sessions of manualized individual CBT for persons meeting DSM-IV-TR diagnostic criteria for GAD. This study will use a treatment manual developed by Dr. Thomas Borkovec and colleagues at the Pennsylvania State University. Participants who meet high endstate functioning criteria and/or achieve remission following CBT will be evaluated periodically during a twenty-four month follow-up phase. Participants who do not meet high endstate functioning criteria and/or achieve remission following completion of CBT will be offered entry into a twelve-week, open-label, flexible-dose trial of escitalopram therapy. Participants receiving escitalopram therapy will be evaluated periodically during a twenty-four month follow-up phase, as well. It is anticipated that patients who do not fully respond to CBT will show a significant increment in improvement in GAD symptoms, over and above their CBT posttreatment level, following pharmacotherapy with escitalopram.

At present, no studies with GAD populations have examined the additive or sequenced effects of psychosocial therapy and SSRI antidepressant pharmacotherapy. The proposed research is a first step in this direction and may provide evidence supporting the use of combined treatment modalities in CBT partial and non-responders.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the ages of 18 and 65 (inclusive)
2. Primary DSM-IV-TR diagnosis of Generalized Anxiety Disorder (GAD) with no significant co-morbid anxiety disorder for which CBT for GAD is not appropriate including PTSD, OCD, and prominent panic disorder with or without agoraphobia
3. A negative urine toxicology, i.e., a urine specimen that does not test positive for use of drugs of abuse, or use of benzodiazepines, in the previous three weeks
4. Penn State Worry Questionnaire score of 55 or greater
5. Have a score of equal to or > 4 (Moderately Ill) on Clinical Global Impression (CGI) Scale (severity of illness item) for GAD
6. Ability to give informed consent
7. Fluent in English
8. Willingness to have Cognitive-Behavioral Therapy sessions audiotaped -

Exclusion Criteria:

1. Patients who have a diagnosis of Major Depressive Disorder within 60 days prior to the clinical interview, and patients who have a "lifetime" history of being diagnosed with one or more of the following disorders: Schizophrenia, Major Depressive Disorder with Psychotic or Catatonic features, Bipolar I Affective Disorder, or Organic Mental Disease
2. DSM-IV substance abuse or dependence within the past 6 months (except nicotine or caffeine)
3. Active suicidal or homicidal ideation, or judged to be at serious suicide risk
4. Hamilton Rating Scale for Depression score of greater than 20 at Screening or Baseline evaluation
5. Any unstable medical or neurological condition
6. Women who are pregnant or lactating
7. Having received CBT treatment for GAD previously
8. Concurrent psychosocial therapy
9. Current psychotropic medication with exception of zolpidem at hs for insomnia
10. History of nonresponse to an adequate trial of escitalopram or intolerable adverse effects to escitalopram -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franklin R. Schneier, M.D., Principal Investigator — New York State Psychiatric Institute; Kenneth D Belzer, Ph.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- Anxiety Disorders Clinic, New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schneier FR, Belzer KD, Kishon R, Amsel L, Simpson HB. Escitalopram for persistent symptoms of generalized anxiety disorder after CBT: a pilot study. J Nerv Ment Dis. 2010 Jun;198(6):458-61. doi: 10.1097/NMD.0b013e3181da4d77. PMID 20531128
- See also: New York State Psychiatric Institute Homepage — http://www.nyspi.org
- See also: Anxiety Disorders Association of America Homepage — http://www.adaa.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive-behavioral Therapy: 14 weekly sessions of individual cognitive-behavioral therapy
Period: Cognitive Behavioral Therapy Phase
Arm/Group | Cognitive-behavioral Therapy
Started | 25
Completed | 15
Not Completed | 10
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 2
Period: Escitalopram Phase
Arm/Group | Cognitive-behavioral Therapy
Started | 7 (7 responders to CBT were ineligible to start and 1 declined, leaving 7 who started escitalopram)
Completed | 4
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Cognitive-behavioral Therapy
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Anxiety Rating Scale Score
Description: The Hamilton Anxiety Rating Scale is a clinician administered rating scale assessing severity of anxiety from 0 (low) to 64 (high). The greater the magnitude of decrease in score during treatment, the greater the improvement in anxiety.
Time Frame: week 14 to week 26
Population: see above: Patients who completed the CBT phase and started escitalopram treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Patients Who Started Escitalopram: Patients who completed the CBT phase and started escitalopram phase treatment
Arm/Group | Patients Who Started Escitalopram
Number analyzed (Participants) | 7
units on a scale | -6.4 (10.1)

2. Primary Outcome: Change in Clinical Global Impressions-Severity Index
Description: 7 point scale of overall severity of psychopathology from 1 mildest to 7 most severe.
Time Frame: week 14 to week 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients Who Started Escitalopram
Number analyzed (Participants) | 7
units on a scale | 1.4 (1.0)

3. Primary Outcome: Change in Generalized Anxiety Disorder Severity Scale
Description: measures severity of symptoms of generalized anxiety disorder, reported as a total score summing 10 items that are each rated from 0, never to 4, all of the time. Range is 0 to 40, with 40 most severe.
Time Frame: week 14 to week 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients Who Started Escitalopram
Number analyzed (Participants) | 7
units on a scale | 4.8 (3.2)

4. Primary Outcome: Change in Penn State Worry Questionnaire
Description: total score (of 16 items) ranging from 16 (least worry) to 80 (most worry)
Time Frame: week 14 to week 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients Who Started Escitalopram
Number analyzed (Participants) | 7
units on a scale | 9.8 (11.2)

5. Primary Outcome: Change in State-Trait Anxiety Inventory, State Subscale
Description: only the total score of the state anxiey subscale was used. Range is from 20 (mildest) to 80 (most severe)
Time Frame: week 14 to week 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients Who Started Escitalopram
Number analyzed (Participants) | 7
units on a scale | 15.4 (11.6)

6. Secondary Outcome: Clinical Global Impressions-Improvement Index
Description: This is a single item rating overall symptomatic improvement. Range is 0 (very much worse) to 7 (very much improved)
Time Frame: week 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients Who Started Escitalopram
Number analyzed (Participants) | 7
units on a scale | 3.0 (1.5)

7. Secondary Outcome: Change in Hamilton Rating Scale for Depression
Description: 24 item version of this standard depression scale, total score ranges from 0 (not depressed) to 58 (most severe)
Time Frame: week 14 to week 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients Who Started Escitalopram
Number analyzed (Participants) | 7
units on a scale | 7.3 (5.9)

8. Secondary Outcome: Change in Beck Depression Inventory-II
Description: total score ranges from 0 (not depressed) to 63 (most severe)
Time Frame: week 14 to week 26
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients Who Started Escitalopram
Number analyzed (Participants) | 7
units on a scale | 10.7 (10.3)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Group 1: all subject entered
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 2/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=25)
insomnia (Nervous system disorders) | 2 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No